CLINICAL TRIAL: NCT07045740
Title: Evaluation of a Novel Role Proposal for the Use of a Physiotherapist Navigator in an Acute Cancer Care Setting in Ontario: a Pilot Randomized Controlled Trial
Brief Title: Physiotherapist Navigator Pilot Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PT Navigator
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PT Navigator (Experimental)
  Interventions: Other: PT Navigator
- Usual Care (No Intervention)

INTERVENTIONS:
Other: PT Navigator — Participants assigned to the intervention group will meet with the PT Navigator withing the first month of starting cancer treatment. Following a one-hour initial assessment, the PT Navigator will follow up every two-three weeks for a total of six sessions. The PT Navigator will administer outcome measures to screen for complications or side effects of treatment. If any complications or side-effects are identified, the PT Navigator will facilitate referrals to other health care practitioners, provide exercise and/or rehabilitation treatment, or provide education and continue monitoring.
  Arms: PT Navigator

SUMMARY:
Background: More Canadians are living with and beyond cancer in Canada. However, most survivors live with harsh side effects due to cancer and its treatments. While international guidelines recommend involving physiotherapists (PTs) in cancer care, many countries do not provide access to these services as a standard part of treatment. Healthcare navigators help patients overcome barriers and streamline care which has shown to improve clinical processes while reducing clinical and patient costs. Through ongoing and routine assessment, a PT Navigator could specifically address issues like fatigue and strength loss, refer patients to other needed services, and help set goals to improve quality of life. Currently, there are no PT Navigator roles in acute cancer care settings in Canada. The purpose of this study is to examine the feasibility and preliminary effectiveness of a PT Navigator role for individuals living with cancer receiving cancer treatment.

Methods:

Participants will include adults recently diagnosed with cancer who are/will be receiving cancer treatment (e.g., chemotherapy, radiation, immunotherapy), are English-speaking and community dwelling. Participants in the intervention group will be followed by the PT Navigator for 12-18 weeks who will screen for early side effects of cancer and its treatment and respond or refer accordingly. Participants in the control group will continue with usual care.

Outcomes: Participants will be assessed at 3 time points. The primary outcome is adherence. Secondary outcomes include other feasibility measures such as retention, recruitment, satisfaction, and preliminary effectiveness will be assessed using overall impairment score, self-reported exercise volume, quality of life, health care utilization, exercise capacity and physical function.

Impact:

If feasible, this will be the first study to facilitate routine PT assessment and early intervention as a component of cancer care in Canada. Findings will inform future methods examining the novel role and can improve the way rehabilitation services are provided to individuals living with or beyond cancer in Canada and internationally.

DETAILED DESCRIPTION:
Rationale: Cancer affects nearly half of Canadians in their lifetime, and while survival rates are improving, many individuals live with long-term side effects that impact their quality of life. Physical activity and rehabilitation have been shown to improve physical function, reduce mental health symptoms, and enhance overall well-being for those living with and beyond cancer. Despite recommendations from international guidelines for physiotherapists (PTs) to be involved in cancer care, only 30% of Canadian cancer survivors have access to rehabilitation services. Incorporating PT Navigators into care teams early into cancer treatment could work to identify and address barriers, provide individualized symptom management, and connect patients with relevant services. However, no research to date has evaluated the role of PTs as navigators in acute cancer care settings in Canada.

Objective and Research Questions:

The objective of this study is to examine the feasibility and preliminary effectiveness of a PT Navigator role for individuals living with cancer receiving cancer treatment (e.g., chemotherapy, radiation, immunotherapy) in an acute cancer care setting.

Research Question 1 (Primary): Is a PT-Navigator role feasible to implement at a cancer institution in Ontario, Canada? Research Question 2 (Secondary): Do individuals with cancer who are monitored by a PT-Navigator demonstrate trends for improved outcomes in overall impairment score, QOL, physical activity levels, exercise capacity, functional strength, activity limitations, and a reduction in health care utilization costs compared to individuals with cancer who are not monitored by a PT Navigator during treatment?

Study Design: Pilot randomized control trial Participants: Adults aged ≥18 years old, recently diagnosed with any type/stage of cancer who are/will be receiving cancer treatment (e.g., chemotherapy, radiation, immunotherapy), English-speaking, and are community-dwelling Procedure: Participants will be randomized to two groups. Intervention Group (PT Navigator): An assessment and 6 follow up sessions approximately every 2-3 weeks with the PT Navigator.

Control Group (Usual Care): No intervention.

Significance:

Results of this study will aim to maximize the success and feasibility of the role when trialed in a future larger scaled randomized controlled trial. The overall goal of the project is to facilitate routine assessment and early intervention as a standard component of cancer care in Canada.

ELIGIBILITY:
Inclusion Criteria:

* adults aged ≥18 years old; recently diagnosed with any type/stage of cancer who are/will be receiving cancer treatment (e.g., chemotherapy, radiation, immunotherapy); English-speaking; are community-dwelling

Exclusion Criteria:

* have a self-reported physical or cognitive impairment that would prevent them from carrying out a physical assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Adherence Rate | 12-18 weeks
  Adherence will be measured dichotomously through attendance (i.e., yes/no) at each session by the PT Navigator

SECONDARY OUTCOMES:
Retention Rate | 12-18 weeks
  Retention will be measured by the number of individuals who complete both a baseline and follow up assessment
Recruitment Rate | 12-18 weeks
  To assess recruitment rate, electronic records will be kept detailing the source and date of recruitment offer and how many eligible referrals are enrolling into the study
Participant Satisfaction | 12-18 weeks
  7-point Likert scale; 1-7 - higher scores indicate greater satisfaction
Participant Satisfaction | 20-26 weeks
  7-point Likert scale; 1-7 - higher scores indicate greater satisfaction
Overall Impairment Score | 12-18 weeks weeks
  Edmonton Symptom Assessment System (ESAS); higher scores represent higher perceived symptom burden; scores ranging from 0 to 10, where 0 indicates the symptom is absent and 10 indicates the worst possible severity
Overall Impairment Score | 20-26 weeks
  Edmonton Symptom Assessment System (ESAS); higher scores represent higher perceived symptom burden; scores ranging from 0 to 10, where 0 indicates the symptom is absent and 10 indicates the worst possible severity
Self-Reported Exercise Volume | 12-18 weeks
  Godin Leisure Time Exercise Questionnaire (higher scores represent higher volume of exercise)
Self-Reported Exercise Volume | 20-26 weeks
  Godin Leisure Time Exercise Questionnaire (higher scores represent higher volume of exercise)
Health-Related Quality of Life | 12-18 weeks
  EORTC QLQ-C30; a high score for a functional scale represents a high level of functioning, a high score for the QoL represents a high QoL, a high score for a symptom scale represents a high level of symptomatology; a scale of 0 to 100
Health-Related Quality of Life | 20-26 weeks
  EORTC QLQ-C30; a high score for a functional scale represents a high level of functioning, a high score for the QoL represents a high QoL, a high score for a symptom scale represents a high level of symptomatology; a scale of 0 to 100
Health-Related Quality of Life | 12-18 weeks
  Functional Assessment of Cancer Therapy - General (FACT-G); higher scores represent better QoL; Total scores range from 0-108
Health-Related Quality of Life | 20-26 weeks
  Functional Assessment of Cancer Therapy - General (FACT-G); higher scores represent better QoL; Total scores range from 0-108
Health Care Utilization | 12-18 weeks
  This questionnaire assesses loss of work, procedures received, and all health-related visits (i.e., family doctor, support services). All costs will be calculated according to current (2025) Ontario healthcare standards and presented in CAD.
Health Care Utilization | 20-26 weeks
  This questionnaire assesses loss of work, procedures received, and all health-related visits (i.e., family doctor, support services). All costs will be calculated according to current (2025) Ontario healthcare standards and presented in CAD.
Physical Functioning | 12-18 weeks
  30 second Sit to Stand
Physical Functioning | 20-26 weeks weeks
  30 second Sit to Stand
Exercise Capacity | 12-18 weeks
  6 minute Walk Test
Exercise Capacity | 20-26 weeks
  6 minute Walk Test

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Smith-Turchyn, PT, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No